CLINICAL TRIAL: NCT04497311
Title: Pulmonary Tomographic Findings in COVID-19 and Influenza H1N1 Patients
Brief Title: Tomographic Findings in COVID-19 and Influenza
Acronym: TOMOCOVIDMX
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universidad de Guanajuato (Other)
Collaborators: Hospital General Regional de León (Other Government); University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Jaime Daniel Mondragón Uribe, Medical researcher, Universidad de Guanajuato
Other Study IDs: HGL-ENSE-00743-20
Record Dates: First submitted 2020-07-31; First posted 2020-08-04 (Actual); Last update posted 2020-08-06 (Actual); Status verified 2020-08

CONDITIONS: SARS-CoV-2; Covid19; H1N1 Influenza; Computed Tomography
Keywords: Radiological patterns; 28-day survival
MeSH Terms: conditions — COVID-19; Orthomyxoviridae Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Nasopharyngeal (NP) specimen, oropharyngeal (OP) specimen, nasal mid-turbinate swab, anterior nares (nasal swab) specimen, nasopharyngeal wash/aspirate or nasal wash/aspirate (NW) specimen or sputum from upper airways.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SARS-CoV-2: Patients with a SARS-CoV-2 polymerase chain reaction positive test upon admission to the emergency department.
  Interventions: Diagnostic Test: Thoraxic computed tomography
- H1N1 influenza: Patients with an influenza H1N1 polymerase chain reaction positive test upon admission to the emergency department.
  Interventions: Diagnostic Test: Thoraxic computed tomography

INTERVENTIONS:
Diagnostic Test: Thoraxic computed tomography — Diagnostic lung CT.

SUMMARY:
The investigators decided to conduct a longitudinal study that compares the pulmonary tomographic patterns found in patients with viral pneumonia (i.e. influenza H1N1 and SARS-CoV-2) at a regional hospital. The primary aim of this study is to compare the radiological patterns found in patients with COVID-19 and influenza H1N1. The secondary aims of this study will assess the association between the radiological CT pattern and the need for invasive mechanical ventilation and mortality within the first 28 days of intensive care unit admission.

DETAILED DESCRIPTION:
Background

In late 2019, a new coronavirus was linked to several cases of pneumonia in the city of Wuhan, Hubei province, China. On February 11, 2020, the World Health Organization (WHO) designated COVID-19 a pandemic disease. The mortality associated with COVID-19 patients that required management in a critical care unit is approximately 4.3%. COVID-19 is caused by severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2). Diagnosis of COVID-19 is made with a positive test (i.e. reverse transcriptase-polymerase chain reaction, RT-PCR) from a person with clinical signs and symptoms of a respiratory tract infection. Viral pneumonia is currently a challenge worldwide as it is associated with high morbidity and mortality. In June of 2009, the WHO declared influenza A H1N1 a pandemic disease. Worldwide, influenza H1N1 had a mortality of 11%, with a higher mortality rate among people older than 50 years of age (i.e. 18-20%). Influenza diagnosis can be established using RT-PCR. Around 200 million cases of community-acquired viral pneumonia occur each year worldwide, 100 million in children, and 100 million in adults. Imaging findings in viral pneumonia are diverse and overlap with findings associated with non-viral infections and inflammatory conditions. However, identifying the underlying viral pathogens may not always be easy. Several imaging patterns have been described in association with these viruses. Although a definitive diagnosis cannot be achieved based on imaging studies, imaging pattern recognition of viral pneumonia can help differentiate between viral and bacterial pathogens; thus, reducing the use of indiscriminate antibiotics. There are few studies that correlate tomographic findings in patients with viral infections in the lower respiratory tract.

The use of computed tomography (CT) should be considered as the first option for diagnostic imaging in patients with suspected pneumonia. Peripheral multifocal ground glass patterns with irregular consolidation images found in the lower lobes or posteriorly in pulmonary CT scans have been described in patients with viral pneumonia due to SARS-CoV-2. Furthermore, complicating the diagnosis of atypical viral pneumonia, 17.9% of mild COVID-19 and 2.9% of moderate-severe COVID-19 patients did not have CT evidence of pneumonia upon hospital admission. One recent study compared the CT radiological patterns found in COVID-19 pneumonia to other viral pneumonias (i.e. influenza, parainfluenza, adenovirus, and respiratory syncytial virus) reporting higher peripheral distribution (i.e. 80% vs. 57%, p<0.001), more ground-glass opacities (i.e. 91% vs 68%, p<0.001), greater frequency of fine reticular opacities (i.e. 56% vs. 22%, p<0.001), and vascular thickening in COVID-19 patients; meanwhile, other viral pneumonias were more likely to have a mixed distribution pattern(i.e. 35% vs. 14%, p<0.001), have pleural effusion (i.e. 39% vs. 4.1%, p<0.001), and present visible lymph nodes (10.2% vs. 2.7%, p<0.001). Another study compared the pulmonary radiological patterns associated with COVID-19 compared to influenza (A and B) reporting higher round opacities (i.e. 35% vs. 17%, p=0.048) and greater frequency of interlobular septal thickening (i.e. 66% vs. 43%, p=0.014) in patients with COVID-19; conversely, influenza patients had a higher frequency of nodular lesions (i.e. 71% vs. 28%, p<0.001), higher frequency of small dense nodular lesions (i.e. 40% vs. 9%, p<0.001), and more likely to have pleural effusion (i.e. 31% vs. 6%, p<0.001).

Research questions

1. What are the pulmonary tomographic findings in patients diagnosed with community-acquired pneumonia secondary to SARS-CoV-2?
2. What are the pulmonary tomographic findings in patients diagnosed with community-acquired pneumonia secondary to H1N1 influenza?
3. Are the 28-day survival distributions different for SARS-CoV-2 and H1N1 influenza?
4. Is there a difference in the 28-day survival distribution and the pulmonary tomographic radiological patterns in patients with pneumonia secondary to SARS-CoV-2?
5. Is there a difference in the 28-day survival distribution and the pulmonary tomographic radiological patterns in patients with pneumonia secondary to H1N1 influenza?
6. What factors are associated with the survival differences in 28-day mortality in both groups and between groups?

ELIGIBILITY:
Inclusion Criteria:

* Patients with signed informed consent.
* Patients with a positive PCR test for SARS-CoV-2 or influenza H1N1 test upon emergency department admission.
* Patients with lung CT within 24hrs of specimen collection for PCR test.
* Patients with complete 30-day follow-up information.

Exclusion Criteria:

* Patients who are unwilling to undergo a lung CT.
* Negative PCR test for SARS-CoV-2 or influenza H1N1 test upon emergency department admission.
* Patients with a tumor or tumor metastasis on the pulmonary CT.
* Patients with a previous or de novo autoimmune disease diagnosis.
* Patients with a previous or de novo interstitial lung disease.
* Pregnancy.

Elimination Criteria:

* Patients with loss of information on the variables of interest.
* Patients without 30-day follow-up information.
* Patients who chose to withdraw their participation at any time of the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Convenience sample from a Mexican urban, suburban, and rural population. The patients come from all demographical and socio-economic strata from a country with a high (0.767) Human Development Index. Our hospital is open to the entire population and primarily assists people with limited to very limited resources.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-06-15 (Actual); Primary Completion 2021-04-30 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
Radiological findings | 24 hours
  Lung CT radiological patterns associated with COVID-19 or Influenza H1N1

SECONDARY OUTCOMES:
Survival | 28 days
  Intrahospital and overall survival at 28 days from hospital admission.

CONTACTS AND LOCATIONS:
Overall Officials: Omar Jiménez-Zarazúa, M.D., Principal Investigator — Medical researcher, Internist
Locations (1):
- Hospital General León-Milenio, León, Guanajuato, Mexico

IPD SHARING:
Plan to Share IPD: Undecided
A database will be generated and available upon request. All patients will de unidentified.

REFERENCES:
- [Result] Wang D, Hu B, Hu C, Zhu F, Liu X, Zhang J, Wang B, Xiang H, Cheng Z, Xiong Y, Zhao Y, Li Y, Wang X, Peng Z. Clinical Characteristics of 138 Hospitalized Patients With 2019 Novel Coronavirus-Infected Pneumonia in Wuhan, China. JAMA. 2020 Mar 17;323(11):1061-1069. doi: 10.1001/jama.2020.1585. PMID 32031570
- [Result] Dandachi D, Rodriguez-Barradas MC. Viral pneumonia: etiologies and treatment. J Investig Med. 2018 Aug;66(6):957-965. doi: 10.1136/jim-2018-000712. Epub 2018 Apr 20. PMID 29680828
- [Result] Fineberg HV. Pandemic preparedness and response--lessons from the H1N1 influenza of 2009. N Engl J Med. 2014 Apr 3;370(14):1335-42. doi: 10.1056/NEJMra1208802. No abstract available. PMID 24693893
- [Result] Louie JK, Acosta M, Winter K, Jean C, Gavali S, Schechter R, Vugia D, Harriman K, Matyas B, Glaser CA, Samuel MC, Rosenberg J, Talarico J, Hatch D; California Pandemic (H1N1) Working Group. Factors associated with death or hospitalization due to pandemic 2009 influenza A(H1N1) infection in California. JAMA. 2009 Nov 4;302(17):1896-902. doi: 10.1001/jama.2009.1583. PMID 19887665
- [Result] Uyeki TM, Bernstein HH, Bradley JS, Englund JA, File TM, Fry AM, Gravenstein S, Hayden FG, Harper SA, Hirshon JM, Ison MG, Johnston BL, Knight SL, McGeer A, Riley LE, Wolfe CR, Alexander PE, Pavia AT. Clinical Practice Guidelines by the Infectious Diseases Society of America: 2018 Update on Diagnosis, Treatment, Chemoprophylaxis, and Institutional Outbreak Management of Seasonal Influenzaa. Clin Infect Dis. 2019 Mar 5;68(6):e1-e47. doi: 10.1093/cid/ciy866. PMID 30566567
- [Result] Ruuskanen O, Lahti E, Jennings LC, Murdoch DR. Viral pneumonia. Lancet. 2011 Apr 9;377(9773):1264-75. doi: 10.1016/S0140-6736(10)61459-6. Epub 2011 Mar 22. PMID 21435708
- [Result] Koo HJ, Lim S, Choe J, Choi SH, Sung H, Do KH. Radiographic and CT Features of Viral Pneumonia. Radiographics. 2018 May-Jun;38(3):719-739. doi: 10.1148/rg.2018170048. PMID 29757717
- [Result] Shiley KT, Van Deerlin VM, Miller WT Jr. Chest CT features of community-acquired respiratory viral infections in adult inpatients with lower respiratory tract infections. J Thorac Imaging. 2010 Feb;25(1):68-75. doi: 10.1097/RTI.0b013e3181b0ba8b. PMID 20160606
- [Result] Upchurch CP, Grijalva CG, Wunderink RG, Williams DJ, Waterer GW, Anderson EJ, Zhu Y, Hart EM, Carroll F, Bramley AM, Jain S, Edwards KM, Self WH. Community-Acquired Pneumonia Visualized on CT Scans but Not Chest Radiographs: Pathogens, Severity, and Clinical Outcomes. Chest. 2018 Mar;153(3):601-610. doi: 10.1016/j.chest.2017.07.035. Epub 2017 Aug 9. PMID 28802696
- [Result] Zu ZY, Jiang MD, Xu PP, Chen W, Ni QQ, Lu GM, Zhang LJ. Coronavirus Disease 2019 (COVID-19): A Perspective from China. Radiology. 2020 Aug;296(2):E15-E25. doi: 10.1148/radiol.2020200490. Epub 2020 Feb 21. PMID 32083985
- [Result] Bai HX, Hsieh B, Xiong Z, Halsey K, Choi JW, Tran TML, Pan I, Shi LB, Wang DC, Mei J, Jiang XL, Zeng QH, Egglin TK, Hu PF, Agarwal S, Xie FF, Li S, Healey T, Atalay MK, Liao WH. Performance of Radiologists in Differentiating COVID-19 from Non-COVID-19 Viral Pneumonia at Chest CT. Radiology. 2020 Aug;296(2):E46-E54. doi: 10.1148/radiol.2020200823. Epub 2020 Mar 10. PMID 32155105
- [Result] Liu M, Zeng W, Wen Y, Zheng Y, Lv F, Xiao K. COVID-19 pneumonia: CT findings of 122 patients and differentiation from influenza pneumonia. Eur Radiol. 2020 Oct;30(10):5463-5469. doi: 10.1007/s00330-020-06928-0. Epub 2020 May 12. PMID 32399710
- [Result] Guan WJ, Ni ZY, Hu Y, Liang WH, Ou CQ, He JX, Liu L, Shan H, Lei CL, Hui DSC, Du B, Li LJ, Zeng G, Yuen KY, Chen RC, Tang CL, Wang T, Chen PY, Xiang J, Li SY, Wang JL, Liang ZJ, Peng YX, Wei L, Liu Y, Hu YH, Peng P, Wang JM, Liu JY, Chen Z, Li G, Zheng ZJ, Qiu SQ, Luo J, Ye CJ, Zhu SY, Zhong NS; China Medical Treatment Expert Group for Covid-19. Clinical Characteristics of Coronavirus Disease 2019 in China. N Engl J Med. 2020 Apr 30;382(18):1708-1720. doi: 10.1056/NEJMoa2002032. Epub 2020 Feb 28. PMID 32109013